CLINICAL TRIAL: NCT01692418
Title: A Randomised Double-blind Controlled Phase III Study to Compare the Efficacy and Safety of Intravenous Ferric Carboxymaltose With Placebo in Patients With Anaemia Undergoing Major Open Abdominal Surgery
Brief Title: Preoperative Intravenous Iron to Treat Anaemia in Major Surgery
Acronym: PREVENTT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12/0246; 2012-002786-35 (EudraCT Number); 10/104/06 (Other Grant/Funding Number: NIHR HTA); 12/EE/0445 (Other: REC); ISRCTN67322816 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2012-09-14; First posted 2012-09-25 (Estimated); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Anaemia
Keywords: Anaemia; Blood transfusion; Surgery; Iron; Ferric carboxymaltose
MeSH Terms: conditions — Anemia | interventions — ferric carboxymaltose; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ferric carboxymaltose (Experimental): 1000mg of ferric carboxymaltose will be administered as an i.v. infusion (100ml normal saline) over a minimum of 15 minutes
  Interventions: Drug: Ferric carboxymaltose; Drug: Normal saline
- Placebo (Placebo Comparator): Normal saline will be administered as an i.v. infusion (100ml normal saline) over a minimum of 15 minutes
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Ferric carboxymaltose — 1000mg of ferric carboxymaltose will be administered as an i.v. infusion (100ml normal saline)
  Other Names: Ferinject
  Arms: Ferric carboxymaltose
Drug: Normal saline — Normal saline will be administered as an i.v. infusion (100ml normal saline)

SUMMARY:
Anaemia is a common problem in patients undergoing surgery. About half of patients undergoing a major operation have anaemia, often a consequence of the disease requiring surgery. Anaemia causes patients to feel tired and unwell. Anaemia at the time of surgery increases the requirement for blood transfusion (50% if anaemic compared to only 15% without anaemia). Both anaemia and blood transfusions are associated with increased complications from surgery, delayed recovery and prolonged hospital stay. The investigators propose that giving intravenous iron before operation can be used to correct anaemia in these patients. Consequently if patients are not anaemic they are less likely to need blood transfusion. Also patients feel better and their health is improved before their operation they are more likely to tolerate the surgery, recover faster, be less likely to have complications from surgery and return home sooner. This will have benefits to the individual patient and also to the NHS by reducing costs.

Oral Iron tablets are not effective as they take 3-6 months to increase blood levels, the tablets are often not tolerated as cause constipation or stomach pain, overall only 30-50% of people continue taking oral iron. A full treatment dose of intravenous iron can be given in 15 minutes with minimal side effects. The effect is to rapidly increase blood counts in 2-4 weeks. The investigators propose that this treatment can be incorporated to patient preparation pathways for surgery as an outpatient without the need for additional visits to hospital.

Small studies have suggested a benefit of iron therapy in orthopaedic and gynaecological surgery. This study will look at 500 patients undergoing major surgery at 20 hospitals in the UK. The investigators anticipate half of patients treated will have their anaemia corrected before operation. Patients with anaemia will be identified as part of the routine blood tests taken preoperatively and invited to take part in the study. Following informed consent, they will be randomly allocated to receive either intravenous iron or a placebo infusion of saline. Intravenous iron is a dark liquid given continuously into a vein over 15 minutes. To ensure neither doctor nor patient knows which treatment is being given both infusions will be prepared and administered by an unblinded authorised person via a black bag through black tubing. There will be no other changes to the patient's normal treatment.

The main aim of this study is to assess if intravenous iron will reduce the need for blood transfusion in the time period around the operation. Further outcome measures will include; patient-reported quality of life, complications, length of hospital stay, and cost. Outcomes will be assessed both during hospital stay and after the patient has been discharged. The trial will be run through a Clinical Trials Unit with considerable experience in conducting large trials. The team has a large range of experience in anaemia management and assessment of complications, quality of life and the cost of health care.

The main aim of this study is to assess if intravenous iron will reduce the need for blood transfusion in the time period around the operation. Further outcome measures will include; patient-reported quality of life, complications, length of hospital stay, and cost. Outcomes will be assessed both during hospital stay and after the patient has been discharged. The trial will be run through a Clinical Trials Unit with considerable experience in conducting large trials. The team has a large range of experience in anaemia management and assessment of complications, quality of life and the cost of health care.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age and signed written informed consent.
2. Patients undergoing elective major open abdominal surgery.

   * The Indication for operation may be for benign or malignant disease.
   * Major Surgery is defined as an operation of anticipated duration more than one hour.
3. Screening haemoglobin (Hb) greater than or equal to 90 g/L (9.0 g/dL) but below or equal to 120 g/L (12.0 g/dL) in women or 130 g/L (13.0 g/dL) in men within four weeks of randomisation.
4. Randomisation and administration of study infusion a minimum of 10 days and maximum 42 days before planned operation.
5. Negative pregnancy test for women of childbearing potential (within last 7 days), and agree to use effective form of contraception until 6 weeks post treatment.
6. Laboratory data used for determination of eligibility at the baseline visit must not be older than four weeks.

Exclusion Criteria:

1. Patients undergoing laparoscopic surgery.
2. Body weight under 50kg.
3. Known history of acquired iron overload, or family history of haemochromatosis or thalassemia or TSAT > 50%.
4. Known reason for anaemia (e.g. untreated B12 or folate deficiency or haemoglobinopathy).
5. Known hypersensitivity to ferric carboxymaltose (Ferinject®) or its excipients.
6. Temperature > 37.5 degrees celsius or patient on non-prophylactic antibiotics
7. Known chronic liver disease
8. If clinically indicated for the patient to have LFT's as part of pre-assessment for surgery and this screening alanine transaminase (ALT) or aspartate transaminase (AST) is above three times the upper limit of the normal range.
9. Received erythropoietin or i.v. iron therapy in the previous 12 weeks.
10. Immunosuppressive therapy (for organ transplantation) or renal dialysis (current or planned within the next 12 months).
11. Patients with severe asthma or severe allergy (requiring hospitalisation within the last 12 months).
12. Unfit for elective surgery.
13. Pregnancy or lactation.
14. Inability to fully comprehend and/or perform study procedures in the investigator's opinion.
15. Patient involvement in another IMP trial within the previous 4 weeks, prior to randomisation. Involvement in another IMP trial, following randomisation, that may impact on the results of the PREVENTT trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 487 (Actual)
Dates: Start 2014-01; Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Risk of blood transfusion or death | From randomisation until 30-days following the index operation
  Co-primary outcome
Blood transfusion rate (including repeat transfusions) | From randomisation until 30-days following the index operation
  Co-primary outcome

SECONDARY OUTCOMES:
Change in haemoglobin levels | From randomisation to (i) day of index operation, (ii) 8-weeks post index operation and (iii) 6 months post index operation
Total number of units of blood or blood products cross matched, total number of packed red cells and any blood products transfused | From randomisation to 30 days post index operation
Post operative morbidity survey (POMS) outcomes (outcomes will be presence of morbidity defined by the domains of the POMS e.g. gastrointestinal, cardiovascular) | At days 3, 5, 7 and 14 following the index operation
Health-related quality of life: Change in The Multidimensional Fatigue Inventory (MFI) questionnaire total score | From baseline to the 10 day assessment and at 8 weeks and 6 months post operatively
Health-related quality of life: Change in European Quality of Life: 5 Dimensions-5 Levels (EQ-5D-5L) questionnaire total score | From baseline to the 10 day assessment and at 8 weeks and six months post operatively
Health-related quality of life: Change in Single Question Outcome Measure (SQOM) | From baseline to the 10 day assessment and at 8 weeks and six months post operatively
Health resource utilisation | Pre-admission, during admission for index operation, 8 weeks post index operation, and 6 months post index operation
Calculated direct, indirect and total costs for the NHS from two perspectives (payer's and societal perspective) | From baseline to 6 months post-surgery
Cost effectiveness of treatment options using relevant effectiveness parameters | From baseline to 6 months post-surgery
Any reaction or side effect from trial therapy
Any reaction or side effect from whole blood or blood product, transfusion reaction
Serious Adverse Events (SAEs) and Suspected Unexpected Serious Adverse Reactions (SUSARs)
Length of hospital stay
Mortality | 8 weeks and 6 months post-operatively
Readmission | Within 8 weeks and within 6 months of the index operation
Blood transfusion | From randomisation to 8 weeks and 6 months post-operatively
Change in e-GFR

CONTACTS AND LOCATIONS:
Overall Officials: Toby Richards, MD FRCS, Principal Investigator — University College, London
Locations (28):
- United Kingdom (28):
  - Basildon University Hospital, Basildon
  - Blackpool Teaching Hospitals, Blackpool
  - Southmead Hospital, Bristol
  - Broomfield Hospital, Broomfield
  - Countess of Chester Hospital, Chester
  - Russells Hall Hospital, Dudley
  - Royal Infirmary of Edinburgh, Edinburgh
  - Queen Elizabeth Hospital, Gateshead
  - Hereford County Hospital, Hereford
  - Hillingdon Hospital, Hillingdon
  - St James's Hospital, Leeds
  - Aintree University Hospital, Liverpool
  - Liverpool Women's Hospital, Liverpool
  - University College London, London
  - Guy's and St Thomas' Hospital, London
  - Imperial College Hospital, London
  - King's College Hospital, London
  - Royal Marsden, London
  - James Cook University Hospital, Middlesbrough
  - Queen's Medical Centre, Nottingham
  - Pennine Acute Hospitals, Oldham
  - John Radcliffe Hospital, Oxford
  - Peterborough and Stamford Hospitals, Peterborough
  - Salford Royal, Salford
  - Northern General Hospital, Sheffield
  - Southampton General Hospital, Southampton
  - Morriston Hospital, Swansea
  - Royal Cornwall Hospital, Truro

REFERENCES:
- [Derived] Richards T, Baikady RR, Clevenger B, Butcher A, Abeysiri S, Chau M, Swinson R, Collier T, Dodd M, Dyck LV, Macdougall I, Murphy G, Browne J, Bradbury A, Klein A. Preoperative intravenous iron for anaemia in elective major open abdominal surgery: the PREVENTT RCT. Health Technol Assess. 2021 Feb;25(11):1-58. doi: 10.3310/hta25110. PMID 33632377
- [Derived] Richards T, Clevenger B, Keidan J, Collier T, Klein AA, Anker SD, Kelly JD. PREVENTT: preoperative intravenous iron to treat anaemia in major surgery: study protocol for a randomised controlled trial. Trials. 2015 Jun 4;16:254. doi: 10.1186/s13063-015-0774-2. PMID 26041028
- See also: Study website — http://preventt.lshtm.ac.uk/